CLINICAL TRIAL: NCT01962324
Title: Phase 2 Study of High Risk Prostatae Cancer Treated With Dose-escalated Simultaneous Integrated Boost to Prostate and Lymph Node GTV
Brief Title: Dose Escalation With SIB to Intraprostatic/Lymphatic GTV in High Risk Prostate Cancer
Acronym: PARAPLY-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Camilla Thellenberg Karlsson, MD, PhD, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARAPLY-1
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Prostatic Neoplasms; Lymphatic Metastasis
Keywords: Quality of Life; Radiotherapy; Radiotherapy, dose-escalation
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SIB Dose-Escalation radiotherapy (Experimental): Simultaneous integrated boost to intraprostatatic tumor and lymph nodes
  Interventions: Radiation: SIB Dose-Escalation Radiotherapy

INTERVENTIONS:
Radiation: SIB Dose-Escalation Radiotherapy

SUMMARY:
A single arm phase 2 study to study the outcome of dose-escalation with simultaneous integrated boost to intraprostatic lesion and positive lymph nodes. Prostate cancer patients with high risk of lymph node metastasis or oligo positive nodes in true pelvic area can be included. The boost volumes will be outlined by usin PET-CT and MRI data. Our hypothesis is that we will have fewer relapses in this very high risk patient group compared to matched historical controls with acceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high risk prostate cancer with a risk of lymphatic spread >15% according to the MSKCC nomogram (1) http://nomograms.mskcc.org/Prostate/PreTreatment.aspx
* Written informed consent
* > 18 years
* Fiducial gold markers implanted in the prostate (min 3)

Exclusion Criteria:

* • Non MR-safe implants or other contraindication to MRI

  * WHO PS>1
  * Previous pelvic irradiation
  * TURP within 6 months
  * IPSS >19
  * Metastatic disease in skeleton, parenchymal organs or lymph nodes outside the pelvis
  * Creatinin clearance < 30ml/min according to http://www.fass.se/LIF/produktfakta/kreatinin.jsp

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
PSA progression free survival | 36 months
  PSA progression defined according to American Society for Therapeutic Radiology and Oncology (ASTRO) Phoenix definition: nadir PSA + 2 ng/mL (on three consecutive measurements with at least one month between each)

SECONDARY OUTCOMES:
Genitourinary Quality of Life | 0 6 12 36 60 months
  Questionnaires distributed to patients at these time intervals regarding side-effects in genitourinary and gastrointestinal domains The questionnaire used is PCSS, Prostate Cancer Symptom Scale The scale goes from 0 to 10 where 0-2 is considered no problems, 3-4 minor problems, 5-7 moderate and 8-10 severe
Gastrointestinal Quality of Life | 0 6 12 36 60 months
  Questionnaires distributed to patients at these time intervals regarding side-effects in genitourinary and gastrointestinal domains The questionnaire used is PCSS, Prostate Cancer Symptom Scale The scale goes from 0 to 10 where 0-2 is considered no problems, 3-4 minor problems, 5-7 moderate and 8-10 severe
Overall Quality of Life | 0 6 12 36 60 months
  Questionnaires distributed to patients at these time intervals regarding side-effects in genitourinary and gastrointestinal domains The questionnaire used is PCSS, Prostate Cancer Symptom Scale The scale goes from 0 to 10 where 0-2 is considered no problems, 3-4 minor problems, 5-7 moderate and 8-10 severe
Sexual Quality of Life | 0 6 12 36 60 months
  Questionnaires distributed to patients at these time intervals regarding side-effects in genitourinary and gastrointestinal domains The questionnaire used is PCSS, Prostate Cancer Symptom Scale The scale goes from 0 to 10 where 0-2 is considered no problems, 3-4 minor problems, 5-7 moderate and 8-10 severe

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Thellenberg Karlsson, MD, Principal Investigator — Umea University
Locations (1):
- Umeå University, Cancercenter, Umeå, Sweden